CLINICAL TRIAL: NCT01746030
Title: Pilot Study of Geriatric Assessments in Senior Adults With Multiple Myeloma
Brief Title: Geriatric Assessments in Senior Adults With Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201207060
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaires: No treatment

SUMMARY:
This study will evaluate the prevalence of geriatric syndromes in older adults with multiple myeloma, examine relationships between baseline geriatrics syndromes and initial treatment selection, and examine risk of functional decline.

Relationship between baseline geriatric questionnaires and initial treatment selection in older adults with newly diagnosed multiple myeloma.

Feasibility of subjects completing the CARG geriatric assessments at baseline, 3 months and 6 months.

Comorbidities or dependence in IADLs at baseline predict decline in functional status at 6 months of follow-up in older adults with newly diagnosed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a diagnosis of multiple myeloma by IMWF criteria: diagnosis must have occurred within 3 months of study enrollment.
* Patient must be ≥ 65 years of age.
* Patient's life expectancy must be ≥ 6 months.
* Patient must be willing to complete follow-up assessments.
* Patient must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patient must not have a diagnosis of smoldering myeloma.
* Patient must not have concomitant amyloidosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Bone Marrow Transplant Clinic at Siteman Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The relationship between initial treatment recommendation and baseline questionnaires assessment | At baseline visit
  The physician caring for the patient will be asked to identify his/her initial treatment recommendations. This includes whether the patient is, in his/her assessment, a candidate for high dose therapy and autologous stem cell transplantation. It will also include whether a 2-drug or 3-drug regimen is recommended initially.

SECONDARY OUTCOMES:
Changes in questionnaires from baseline to 6 months | Through 6 months of follow-up
  Logistic regression analyses, adjusted odds ratios (ORs) based on model will be given with 95% CIs. All analyses will use two-tailed significance levels of 0.05 and will be conducted with statistical software SAS 9.2. Geriatric assessment variables will be analyzed as continuous or ordinal variables as indicated. Candidate variables will include: demographic data (including age, gender, race), disease data (stage, cytogenetic abnormalities), or geriatric assessment variables (comorbidity, functional status, physical function, psychological state, nutrition, social support and social activity). Analyses will be performed for the outcomes of treatment selection (transplant vs non-transplant) and increased dependence in IADLs
Completion of the questionnaires at baseline, 3 months and 6 months. | Baseline, 3 months, and 6 months
  Feasibility of subjects completing questionnaires is defined as 90% of consenting subjects completing the baseline geriatric assessment battery, and 80% of consenting subjects completing follow-up assessments at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Wildes, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu